CLINICAL TRIAL: NCT07293000
Title: Evaluation of the Effectiveness of Two Different Nursing Interventions in Preventing Urinary Retention in Patients Undergoing Spinal Anesthesia: Randomized Controlled Trial
Brief Title: Evaluating Two Nursing Interventions to Prevent Urinary Retention After Spinal Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Hülya CEYHAN, Principal Investigator Phd candidate of nursing, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HCEYHAN
Record Dates: First submitted 2025-12-07; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Urinary Retention; Urinary Retention
Keywords: Urinary retention; Postoperative urinary retention; Nursing Interventions; Bladder Volume Measurement Device; Cold Application; Sacral Massage
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, three-arm trial comparing suprapubic cold pack application, sacral massage, and usual care in adults undergoing scrotal, inguinal, pelvic, lower abdominal, or orthopedic surgery with spinal anesthesia.
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomly assigned to one of three groups using a computer-generated random sequence (Randomizer.org), with group allocation concealed in sealed opaque envelopes until enrollment. All interventions will be delivered by a single nurse researcher, who will be aware of group assignments. However, the data will be analyzed by an independent expert who will be blinded to group allocation and will work with de-identified, coded data only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Suprapubic Cold Pack Group (Experimental): Participants in this arm receive a suprapubic dry cold pack in addition to usual postoperative nursing care after surgery with spinal anesthesia. The cold pack is applied in the early postoperative period according to a standard nursing protocol.
  Interventions: Other: Suprapubic Cold Pack
- Sacral Massage Group (Experimental): Participants in this arm receive sacral massage in addition to usual postoperative nursing care after surgery with spinal anesthesia. The massage is delivered in the early postoperative period by a nurse researcher following a standard nursing protocol.
  Interventions: Other: Sacral Massage
- Usual Care Control Group (No Intervention): Participants in this arm receive only usual postoperative nursing care after surgery with spinal anesthesia, according to the hospital's standard protocols. They do not receive any additional study-specific intervention.

INTERVENTIONS:
Other: Suprapubic Cold Pack — A dry cold pack applied externally to the skin over the lower abdomen above the bladder (suprapubic area) in adult patients after surgery with spinal anesthesia. The cold pack is used for a predefined duration in the early postoperative period as a non-pharmacologic, non-invasive nursing intervention to support bladder emptying and patient comfort.
  Arms: Suprapubic Cold Pack Group
Other: Sacral Massage — A gentle manual massage applied externally to the skin over the lower back in the sacral (tailbone) region in adult patients after surgery with spinal anesthesia. The massage is performed for a predefined duration in the early postoperative period as a non-pharmacologic, non-invasive nursing intervention to support bladder function and patient comfort.
  Arms: Sacral Massage Group

SUMMARY:
The goal of this clinical trial is to learn whether two simple nursing methods can help prevent trouble emptying the bladder (acute urinary retention, AUR) after surgery with numbing medicine in the lower back (spinal anesthesia). Adults having surgery in the scrotum (scrotal), groin (inguinal), pelvic area, lower belly (lower abdominal), or bones and joints (orthopedic surgery) with spinal anesthesia will take part. After surgery, participants will be randomly placed into one of three groups: one group will receive a cold pack on the lower belly (suprapubic area), a second group will receive a gentle massage on the lower back over the tailbone (sacral area), and a third group will receive usual care only with no extra procedure. The same nurse researcher will provide the study care for all groups, check how well participants pass urine, use a small painless scan on the lower belly to see how much urine is in the bladder (portable bladder ultrasound), and record whether a tube in the bladder to drain urine (urinary catheter) is needed.

DETAILED DESCRIPTION:
Trouble emptying the bladder after surgery (acute urinary retention, AUR) is a common and important problem in adults who receive numbing medicine in the lower back (spinal anesthesia). AUR can cause pain, an overfilled bladder (bladder distension), urinary tract infection, longer hospital stays, and higher health care costs. The usual way to manage AUR is to place a tube into the bladder to drain urine (urinary catheterization). This works, but it is invasive and may lead to infection, injury to the urethra, and discomfort. Because of these risks, there is a need for simple, non-drug, non-invasive nursing methods to help prevent AUR.

Spinal anesthesia can temporarily block normal bladder function and increase the risk of AUR. Nurses are often the first to notice when a person is unable to pass urine and are in a key position to provide early, preventive care. Some studies have looked at different nursing interventions for urinary retention, but there is little evidence about non-invasive methods after spinal anesthesia, and no trial has directly compared a cold pack on the lower belly with a massage over the tailbone in this setting.

This randomized controlled trial will include adult surgical patients who receive spinal anesthesia for operations in the scrotum (scrotal), groin (inguinal), pelvic area, lower belly (lower abdominal), or bones and joints (orthopedic surgery). Participants will be randomly assigned to one of three groups:

1. a dry cold pack applied to the lower belly over the bladder (suprapubic area),
2. gentle massage over the lower back in the area of the tailbone (sacral area), or
3. usual postoperative care without an extra study procedure.

All study procedures in all three groups will be carried out by a single nurse researcher, using the same assessment steps for every participant. The aim is to keep the care consistent and reduce differences that are not related to the study methods.

The main focus of the study is to find out whether these nursing methods can lower the rate of acute urinary retention after spinal anesthesia. Nurses will regularly check how well participants can pass urine on their own and will estimate bladder volume using a small, painless scan placed on the skin over the lower belly (portable bladder ultrasound device). This objective measurement is expected to improve early detection of AUR compared with relying only on symptoms or physical examination.

The study will also look at related outcomes such as time to first spontaneous urination, need for urinary catheterization, bladder fullness and pain, and comfort and satisfaction with nursing care. By providing clear, comparative information on two simple, non-invasive nursing interventions, this trial aims to support evidence-based postoperative nursing protocols, improve patient comfort, and reduce the need for invasive urinary catheterization after spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria: Patients who meet all of the following criteria will be included:

* Age 18 years or older
* No diagnosis of urolithiasis, benign prostatic hyperplasia, neurogenic bladder, cancer, or other malignancy
* No diagnosis of urinary tract infection within the last month
* No history of prior urological surgery or surgery involving the sacral region
* No history of urinary retention
* Not using antidepressants, antipsychotics, muscarinic receptor antagonists, alpha-blockers, or similar medications
* No contraindication for applying cold to the suprapubic area or massage to the sacral area (e.g., no pacemaker, bladder stimulator, or other sensitive electronic medical device in the sacral region)
* No visual, hearing, cognitive, or perceptual impairment

Exclusion Criteria:Patients who meet any of the following criteria will be excluded:

* Duration of surgery longer than 2 hours
* Urinary catheterization performed preoperatively, intraoperatively, or postoperatively
* Blood transfusion performed preoperatively, intraoperatively, or postoperatively
* Development of complications such as hypothermia, bleeding, or other conditions that prevent the application of dry cold or sacral massage in the preoperative, intraoperative, or postoperative period
* Transfer to the intensive care unit after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Acute Urinary Retention | Postoperative 0-6 hours after surgery with spinal anesthesia
  Proportion of participants who develop postoperative acute urinary retention (AUR) within the first 6 hours after surgery with spinal anesthesia, defined as inability to void spontaneously requiring urinary catheterization and/or elevated bladder volume on bladder ultrasound.

SECONDARY OUTCOMES:
Need for Urinary Catheterization Within the First 6 Hours | Within the first 6 hours after surgery with spinal anesthesia (postoperative 0-6 hours)
  Proportion of participants who require insertion of a urinary catheter due to inability to void or clinically significant bladder distension within the first 6 hours after surgery with spinal anesthesia.
Bladder-Related Discomfort/Pain Score During the First 6 Hours | Within the first 6 hours after surgery with spinal anesthesia (postoperative 0-6 hours)
  Bladder-related discomfort or pain intensity assessed using a numerical rating scale (0-10) during the first 6 hours after surgery with spinal anesthesia
Time to First Spontaneous Voiding Within the First 6 Hours | Within the first 6 hours after surgery with spinal anesthesia (postoperative 0-6 hours)
  Elapsed time in minutes from the end of surgery with spinal anesthesia to the first spontaneous urination without urinary catheterization, measured during the first 6 postoperative hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Institute of Graduate Studies, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://lisansustuegitim.iuc.edu.tr/tr/_